CLINICAL TRIAL: NCT04919122
Title: Outcomes Database to prospectivelY aSSEss the Changing TherapY Landscape in Renal Cell Carcinoma (ODYSSEY RCC)
Brief Title: Outcomes Database to prospectivelY aSSEss the Changing TherapY Landscape in Renal Cell Carcinoma
Acronym: ODYSSEY RCC
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other); Bristol-Myers Squibb (Industry); Exelixis (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00107408
Record Dates: First submitted 2021-05-24; First posted 2021-06-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: ODYSSEY; mRCC; Metastatic Renal Cell Carcinoma; RCC; PRO
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 36.5 mL of blood will be collected within (≤) 3 months of enrollment. Patients only receive a blood draw at their enrollment visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with mRCC with ≤ 3 mos of 1L or 2L systemic therapy: This is an observational cohort.
  * mRCC = metastatic renal cell cancer
  * 1L=first-line systemic therapy
  * 2L=second-line systemic therapy

SUMMARY:
ODYSSEY RCC is a prospective, observational Phase IV study is to understand the cancer management and health-related quality of life in patients with mRCC in routine real-world clinical practice in the United States, including both community and academic treatment settings.

DETAILED DESCRIPTION:
This trial is a prospective, observational Phase IV study is to understand the cancer management and health-related quality of life in patients with mRCC in routine real-world clinical practice in the United States, including both community and academic treatment settings. Primarily, the study will evaluate patient experience through collection of patient reported outcomes (PROs). The study will also collect and assess information on the therapies used such as first-line treatment selection, treatment sequence and duration, the drivers of physician selection of particular agents, and discontinuation of therapies.

The primary objective is to determine distinct patterns of change in the quality of life and symptom burden in mRCC patients receiving therapy.

Patients will be identified and undergo consent and baseline assessments, including research blood collection and processing, by the study site team, this baseline visit will be their only clinic visits per protocol. All other visits are standard of care visits and outside the scope of the study.

Subsequent follow up with be coordinated centrally by DCRI. Additional clinic data will be obtained via PCORnet data pull and Medicare claims. Patient reported outcomes, quality of life and medications data will be obtained via the DCRI Call Center through follow-up phone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or over at time of informed consent.
* Diagnosis of metastatic renal cell cancer (mRCC) with less than or equal to (≤) 3 months of first-line systemic therapy or less than or equal to (≤) 3 months of second-line systemic therapy for mRCC.

  1. Prior surgery and radiation therapy are permitted.
  2. Prior neoadjuvant and adjuvant therapy for non-metastatic renal cell carcinoma are permitted.
  3. Patients currently not on therapy and being observed are permitted.
* Evidence of signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
* Ability to comply with completion of PROs

Exclusion Criteria:

* Patients being treated for metastatic solid tumors other than mRCC are excluded. Non-cytotoxic oral agents for adjuvant or maintenance therapy of other cancers are permitted.
* Patients who are not intending to undergo follow up care at a study site within PCORnet

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic renal cell cancer (mRCC) will be identified and undergo consent and baseline assessments, including research blood collection and processing. Patient reported outcomes will be collected at baseline (pre-treatment) every 3 months for 2 years, and then every 6 months until end of follow up (with a minimum follow-up of 18 months and a maximum follow-up period of 36 months; additional follow up will be obtained based on continuous funding).
Sampling Method: Probability Sample
Enrollment: 468 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in medication adherence as measured by patient report. | baseline, every 3 months for 2 years, every 6 months for up to 36 months
  Patient's report their medication at each study visit.
Change in quality of life in mRCC patients receiving therapy as measured by FKSI-19 | baseline, every 3 months for 2 years, every 6 months for up to 36 months
  The FKSI-19 is a questionnaire about the disease-related symptoms - physical, disease-related symptoms - emotional, treatment side-effects, and function/well-being.
Change in symptom burden in mRCC patients receiving therapy as measured by FKSI-19 | baseline, every 3 months for 2 years, every 6 months for up to 36 months
  The FKSI-19 is a questionnaire about the disease-related symptoms - physical, disease-related symptoms - emotional, treatment side-effects, and function/well-being.
Change in quality of life in mRCC patients receiving therapy as measured by FACT-G | baseline, every 3 months for 2 years, every 6 months for up to 36 months
  The FACT-G is a questionnaire about the physical well-being, social/family well-being, emotional well-being, and functional well-being.
Change in symptom burden in mRCC patients receiving therapy as measured by FACT-G | baseline, every 3 months for 2 years, every 6 months for up to 36 months
  The FACT-G is a questionnaire about the physical well-being, social/family well-being, emotional well-being, and functional well-being.

SECONDARY OUTCOMES:
First line management choice(s) | Up to 36 months
  A composite of REDCap data entry by sites, PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on line management choice(s).
Subsequent line management choice(s) | Up to 36 months
  A composite of REDCap data entry by sites, PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on line management choice(s).
Dosing (starting dose, dose intensity, ending dose) | Up to 36 months
  A composite of REDCap data entry by sites, PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on dosing.
Dose holds and dose interruptions | Up to 36 months
  A composite of PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on dosing holds and interruptions.
Time on treatment | Up to 36 months
  A composite of REDCap data entry by sites, PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on time on treatment.
Time to next treatment | Up to 36 months
  A composite of PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on time to next treatment.
Early discontinuation of one agent of a combination | Up to 36 months
  A composite of PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on early discontinuation of one agent of a combination.
Concomitant glucocorticoid use | Up to 36 months
  A composite of PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on concomitant glucocorticoid use.
Work Productivity and Activity Impairment (WAPI) questionnaire | Up to 36 months
  A composite of REDCap data entry by sites, PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on the WAPI questionnaire.
Health care resource utilization (including hospitalizations) | Up to 36 months
  A composite of PCORnet data pull, Medicare data pull, Physician questionnaire and patient follow-up interviews will be used to get data on health care resource utilization.
Overall survival (OS) of mRCC patients | Up to 36 months
  A composite of various starting points (time of diagnosis of metastatic disease, time of study entry and time of starting systemic therapy) to avoid lead-time bias.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (14):
- United States (14):
  - State University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation d/b/a Ochsner Health, New Orleans, Louisiana
  - The Johns Hopkins University, Baltimore, Maryland
  - The Regents of the University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhavsar NA, Harrison MR, Scales CD, Zhang T, Troy J, Ward K, Jabusch SM, Lampron Z, George DJ. Design and Rationale of the Outcomes Database to Prospectively Assess the Changing Therapy Landscape in Renal Cell Carcinoma Registry: A Multi-institutional, Prospective Study of Patients with Metastatic Renal Cell Carcinoma. Eur Urol Open Sci. 2024 Jul 3;66:75-81. doi: 10.1016/j.euros.2024.06.007. eCollection 2024 Aug. PMID 39070100
- [Derived] Ged Y, Markowski MC, Singla N, Rowe SP. The shifting treatment paradigm of metastatic renal cell carcinoma. Nat Rev Urol. 2022 Nov;19(11):631-632. doi: 10.1038/s41585-022-00651-9. PMID 36064785